CLINICAL TRIAL: NCT05752903
Title: Comparison Between Dexmedetomidine-Propofol and Ketamine-Propofol Administration for Sedation of CT Guided Bone Biopsy: A Randomized Controlled Trial
Brief Title: Dexmedetomidine-Propofol Versus Ketamine-Propofol for Sedation of CT Guided Bone Biopsy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AP2207-50109
Record Dates: First submitted 2023-02-21; First posted 2023-03-03 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-03

CONDITIONS: Sedation
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine-propofol (Active Comparator): Dexmedetomidine-propofol bolus will be administered then Dexmedetomidine-propofol infusion continued during the procedure
  Interventions: Drug: Dexmedetomidine-propofol
- ketamine-propofol (Active Comparator): ketamine-propofol bolus will be administered then Dexmedetomidine-propofol infusion continued during the procedure
  Interventions: Drug: Ketamine-Propofol

INTERVENTIONS:
Drug: Dexmedetomidine-propofol — 1 microgram/kg dexmedetomidine+2.5 mg/kg propofol intravenous (IV) bolus, 0.5 microgram g/kg/h dexmedetomidine+2.5 mg/kg/h propofol infusion
  Other Names: precedex
  Arms: Dexmedetomidine-propofol
Drug: Ketamine-Propofol — 1 mg/kg ketamine+2.5 mg/kg propofol iv bolus, 0.25 mg/kg/h ketamine+2.5mg/kg/h propofol infusion
  Other Names: ketofol
  Arms: ketamine-propofol

SUMMARY:
This study aims to compare the effectiveness and safety of a dexmedetomidine-propofol combination and a ketamine-Propofol combination for sedation of CT guided bone biopsy.

DETAILED DESCRIPTION:
Assessment of boney lesions is an common activity in the care of cancer patients. CT guided Percutaneous needle biopsies have a low complication rate. usually, this procedure is done under sedation.

Propofol is a non-barbiturate hypnotic and sedative. It facilitates gamma-aminobutyric acid mediated inhibitory neurotransmission. It's known to have anti-emetic, antipruritic, anticonvulsant and amnestic effects. Despite being effective and potent, Propofol's main disadvantages is its dose-dependent hypotension and respiratory depression .Ketamine is a phencyclidine derivative which acts as a N-methyl-D-aspartate (NMDA) receptor antagonist. It is a dissociative anesthetic and provides some analgesia. It maintains airway reflexes and spontaneous respiration. Combining Propofol and ketamine preserves the sedative and analgesic efficacy while reducing their adverse effects. Dexmedetomidine is a highly selective α2-agonist. It is eight times more specific compared with clonidine. It has a perioperative anxiolytic, sedative properties as well as some analgesic properties .Dexmedetomidine is usually used for mild to moderate sedation and Propofol could be added to deepen the level of sedation

ELIGIBILITY:
Inclusion Criteria:

* Stated willingness to comply with all study procedures and availability for the duration of the study .
* Age between 18 to 60 years old
* American Society of Anesthesiologists (ASA) physical I-III
* Scheduled for CT guided bone biopsy with sedation.

Exclusion Criteria:

* Severe heart, lung, and liver disease
* kidney failure
* Bleeding diathesis Allergy to drugs to be used

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-03-04 (Actual); Primary Completion 2023-09-10 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Heart rate | before administration (baseline), every 10 minutes during the procedure, every 15 minutes for one hour postoperatively
  change in heart rate

SECONDARY OUTCOMES:
Mean arterial blood pressure | before administration (baseline), every 10 minutes during the procedure, every 15 minutes for one hour postoperatively
  change in the mean arterial blood pressure
Visual analogue scale (VAS) score for pain | every 15 minutes for one hour postoperatively
  assessment of postoperative pain using the visual analogue scale score. the scale is a straight horizontal line (100 mm). The ends are defined as the extreme limits of pain orientated from the left (no pain) to the right (worst pain).The patient marks on the line the point that they feel represents their perception of their current state.
  The VAS score is determined by measuring in millimetres from the left hand end of the line to the point that the patient marks.higher VAS score means worse pain
recovery time | immediately postoperative
  recovery time

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Salah abdelgalil, MD, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National cancer institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No